CLINICAL TRIAL: NCT07142395
Title: Comparison of Primary Skin Closure Versus Delayed Primary Skin Closure in Patients Undergoing Emergency Laparotomies
Brief Title: Comparing Delayed vs Primary Wound Closure After Emergency Laparotomy: Impact on Infection, Healing, and Hospital Stay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bkahtawar Amin Medical and Dental College Multan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1326-2839
Record Dates: First submitted 2025-08-06; First posted 2025-08-26 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Laparotomy Closure After Abdominal Surgery
Keywords: wound infection; primary wound closure; delayed wound closure; Wound dehiscence
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Closure (Active Comparator): Skin closed immediately after laparotomy
  Interventions: Procedure: Immediate skin closure
- Delayed Primary Closure (Experimental): Skin closed 3 - 5 days after laparotomy
  Interventions: Procedure: Delayed primary closure

INTERVENTIONS:
Procedure: Immediate skin closure — After laparotomy wounds will be closed primarily using no. 1 vicryl suture
  Arms: Primary Closure
Procedure: Delayed primary closure — Deeper layers of wound will be closed after surgery and loose mattress sutures will be applied to skin with prolene. After three to five days of daily dressing with bactericidal solution, the skin will be closed
  Arms: Delayed Primary Closure

SUMMARY:
The purpose of this study is to find out which type of wound closure after emergency abdominal surgery leads to fewer wound infections and better recovery: closing the wound immediately after surgery (called primary closure) or waiting a few days before closing the skin (called delayed primary closure).

Wound infection is a common problem after emergency abdominal surgery (also called laparotomy). Some surgeons close the skin right away, while others wait a few days to reduce the risk of infection.

This study will help find out which method is better.

The main questions the study aims to answer are:

1. . Does delayed primary closure lower the rate of wound infection compared to primary closure?
2. . Does the wound open up (wound dehiscence) less often with delayed closure?
3. . Does delayed closure affect the length of hospital stay?

In this clinical trial:

* Adult patients needing emergency abdominal surgery will be included.
* Half the patients will have their wounds closed immediately (primary closure), and half will have delayed closure after 3-5 days of daily dressing.
* All surgeries will be done by experienced surgeons using the same technique.
* Patients will be followed for 4 weeks after surgery to monitor wound infection, wound opening, and length of hospital stay.

The results will help doctors choose the safest and most effective way to close surgical wounds after emergency abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 - 60 years of age
* Either male or female gender and
* Planned to undergo emergency laparotomy

Exclusion Criteria:

* Patients undergoing second laparotomy
* Re- laparotomy
* On steroid therapy and
* Patients who die within 28-days of surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Wound Infection | From date of surgery to Four weeks postoperatively
  Surgical Site infection - Presence any features of erythema, pain, pus discharge on examination of surgical wound and new onset fever (> 98.6 F)

OTHER OUTCOMES:
Hospital Stay | From date of surgery until date of hospital discharge, up to 28 days
  Duration of stay (days) in hospital after laparotomy
Wound dehiscence | From date of laparotomy to Four weeks post-operatively
  A partial or total separation of previously approximated wound edges

CONTACTS AND LOCATIONS:
Overall Officials: Amjad A Professor, FRCS, Study Chair — Bakhtawar Amin Medical and Dental College
Locations (1):
- Bakhtawar Amin Medical and Dental College, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No